CLINICAL TRIAL: NCT03818685
Title: A Multicenter, Randomised, Open-label Phase II Study to Evaluate the Clinical Benefit of a Post-operative Treatment Associating Radiotherapy + Nivolumab + Ipilimumab Versus Radiotherapy + Capecitabine for Triple Negative Breast Cancer Patients With Residual Disease After Neoadjuvant Chemotherapy
Brief Title: Evaluate the Clinical Benefit of a Post-operative Treatment Associating Radiotherapy + Nivolumab + Ipilimumab Versus Radiotherapy + Capecitabine for Triple Negative Breast Cancer Patients With Residual Disease
Acronym: BreastImmune03
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ET17-093 BreastImmune03
Record Dates: First submitted 2019-01-18; First posted 2019-01-28 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer; Triple Negative Breast Neoplasms
Keywords: Residual disease with RCB of Class II or III
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Nivolumab; Ipilimumab; Capecitabine

STUDY DESIGN:
Intervention Model Description: This trial is an open-label, randomised, multicentric, comparative, Phase II study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nivolumab + Ipilimumab (Experimental): Nivolumab (360 mg IV, every 3 weeks) for 8 doses and Ipilimumab (1 mg/kg, IV, every 6 weeks or every 2 doses of Nivolumab in case of dose delays) for 4 doses.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- Capecitabine (Active Comparator): Capecitabine (1000 mg/m2 twice a day, Bis In Die), 14 days on / 7 days off for 8 cycles.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Nivolumab — Radiotherapy will be maintained in each Arm.
  Arms: Nivolumab + Ipilimumab
Drug: Ipilimumab — Radiotherapy will be maintained in each Arm.
  Arms: Nivolumab + Ipilimumab
Drug: Capecitabine — Radiotherapy will be maintained in each Arm.
  Arms: Capecitabine

SUMMARY:
To evaluate the clinical benefit of a post-operative adjuvant therapy combining radiotherapy + Nivolumab + Ipilimumab versus radiotherapy + Capecitabine in Triple Negative Breast Cancer (TNBC) patients with residual disease after neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
This trial is an open-label, randomised, multicentric, comparative, Phase II study aiming to evaluate the clinical benefit of a combined treatment associating radiotherapy + Nivolumab + Ipilimumab versus radiotherapy + Capecitabine (standard treatment) in early TNBC patients who have Residual cancer burden (RCB) II or III residual disease after neoadjuvant chemotherapy.

Following validation of eligibility criteria, patients will be randomised (1:1) to receive:

* Arm A: Nivolumab (360 mg IV, every 3 weeks) for 8 doses and Ipilimumab (1 mg/kg, IV, every 6 weeks or every 2 doses of Nivolumab in case of dose delays) for 4 doses.
* Arm B: Capecitabine (1000 mg/m2 twice a day, Bis In Die [BID]), 14 days on / 7 days off for 8 cycles.

In both arms, radiotherapy will be administered as per standard practice and has to be initiated one week before C1D1.

ELIGIBILITY:
Inclusion Criteria:

* Female patient 18 years of age on day of signing informed consent form.
* Histologically proven TNBC defined as follows : HER2 negativity must be confirmed (by one of the following: Fluorescence in situ hybridization (FISH) negative (FISH ratio <2.2), or Immunohistochemistry (IHC): 0-1+, or IHC 2-3+ and FISH-negative (FISH ratio <2.2)) and less than 1% of cells stained by immunohistochemistry (IHC) for ER and PR as per ASCO guidelines.
* TNBC previously treated by : Standard neoadjuvant chemotherapy containing anthracycline and taxanes and Surgery.
* TNBC patients currently treated by post-operative radiotherapy as per standard and/or institutional guidelines.
* No radiological evidence of metastatic disease documented by a CT-Scan of Chest abdomen and pelvis.
* Residual disease with RCB of Class II or III documented before randomisation using the surgery specimen.
* Availability of a representative formalin-fixed paraffin-embedded (FFPE) tumor block from surgery specimen with its histological report.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1.
* Adequate end organ and bone marrow function as defined in protocol. All screening lab tests should be performed within 7 days before C1D1.
* Absence of significant treatment-related toxicity i.e. > Grade 1 as per CTCAE v5.0, except alopecia (all grades are acceptable), neuropathy (Grade 2 is acceptable) or biological values as defined in protocol.
* Minimal wash-out period for prior treatments (i.e. minimal delay from last dose of prior treatment to C1D1): any investigational agent > 4 weeks (or 5 half-lives whichever is longer with a minimum of 2 weeks), any monoclonal antibody > 4 weeks, any targeted therapies > 4 weeks, - live vaccine > 4 weeks, systemic steroids at doses higher than 10 mg/day prednisone equivalent or other immunosuppressive agents > 3 weeks, sorivudine or its chemically related analogues such as brivudine > 4 weeks.
* Women of child-bearing potential must have a negative serum pregnancy test within 7 days before C1D1.
* Women of child-bearing potential must agree to use 1 effective form of contraception from the time of the negative pregnancy test up to 5 months after the last dose of study drugs.
* Patient should understand, sign, and date the written voluntary informed consent form at the screening visit prior to any protocol-specific procedures performed.
* Patient should be able and willing to comply with study visits and procedures as per protocol.
* Patients must be covered by a medical insurance.

Exclusion Criteria:

* Patient has a metastatic TN breast cancer.
* Patient has previously received therapy with an anti- PD-1, anti- PD-L1, or anti-CTLA4 or any other immunotherapies.
* Patient has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone curative therapy and other completely treated prior malignancy if no evidence of disease for ≥ 2 years.
* Patient presents a contraindication to Nivolumab or Ipilimumab treatment as per respective SPC including known hypersensitivity to one of these study drugs or severe hypersensitivity reaction to any monoclonal antibody.
* Patient presents a contraindication to Capecitabine treatment as per SPC including : 1) History of severe and unexpected reactions to fluoropyrimidine therapy, 2) Hypersensitivity to Capecitabine or to any of the excipients listed in SPC or fluorouracil, 3) Patients with known complete absence of dihydropyrimidine dehydrogenase activity, 4) Treatment with sorivudine or its chemically related analogues, such as brivudine, 5) any contraindication listed in respective SPC.
* Patient has active autoimmune disease that has required systemic treatment in the past 3 months before C1D1 or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids at doses higher than 10 mg/d prednisone equivalents or immunosuppressive agents.
* Patient requires the use of one of the following forbidden treatment during the study treatment period: any investigational anticancer therapy other than the protocol specified thérapies, any concurrent chemotherapy, immunotherapy, biologic for cancer treatment, other than the ones stated in the protocol. Concurrent use of hormones for non-cancer-related conditions (e.g., insulin for diabetes and hormone replacement therapy) is acceptable, major surger, live vaccines, immunosuppressive agents and immunosuppressive high doses of systemic corticosteroids i.e. doses >10 mg/d prednisone or equivalent, sorivudine or its chemically related analogues such as brivudine and any treatment contra-indicated as per Capecitabine SPC.
* History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e. bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan.
* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within 3 months prior to C1D1 unstable arrhythmias or unstable angina, Known Left Ventricular Ejection Fraction (LVEF) < 50%.
* Patient has a known history of active Bacillus Tuberculosis.
* Patient has an active infection requiring systemic therapy.
* Patient has Active hepatitis B (chronic or acute; defined as having a positive hepatitis B surface antigen [HBsAg] test at screening), Active hepatitis C (Patients positive for hepatitis C virus (HCV) antibody are eligible only if PCR is negative for HCV RNA at screening) or Human Immunodeficiency Virus (HIV) infection (HIV 1/2 antibodies).
* Prior allogeneic bone marrow transplantation or solid organ transplant in the past.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive children within the projected duration of the trial, starting with the screening visit through 5 months after the last dose of study drugs.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) | At 2 years
  DFS is defined as the time from randomization until the date of the first relapse (local/regional recurrence or distant metastasis) or death (from any cause) whichever comes firsts and regardless of whether the patient withdraws from randomised study treatment or receives another anti-cancer therapy prior to disease relapse.

SECONDARY OUTCOMES:
Overall survival | Up to 2 years
  Overall survival will be measured from the date of randomization to the date of death from any cause.
Local-regional recurrence | Up to 2 years
  Local-regional recurrence (LRR) refers to relapse of the primary tumor site
Distant metastasis | Up to 2 years
  Distant metastasis is defined as presence of any non-local metastatic sites.
Disease recurrence/relapse (local or distant) | Up to 2 years
  Rate of patients with recurrence at 1 year and 2 year post-randomisation as well as time to recurrence will be analysed.
Adverse Event | Up to 2 years
  The assessment of safety will be based mainly on the frequency of adverse events based on the common toxicity criteria (CTCAE-V5.0) grade.
EORTC QLQ C30 | At Baseline, every 12 weeks and 30 days after the last dose
  Patient reported outcomes and quality of life will be assessed using the validated following questionnaire: The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ C30). The QLQ-C30 incorporates nine multi-item scales: five functional scales (physical, role, cognitive, emotional, and social); three symptom scales (fatigue, pain, and nausea and vomiting); and a global health and quality-of-life scale. Several single-item symptom measures are also included. See scoring manual at :https://www.eortc.be/qol/files/SCManualQLQ-C30.pdf.
Questionnaire EORTC QLQ BR-23 | At Baseline, every 12 weeks and 30 days after the last dose
  Patient reported outcomes and quality of life will be assessed using the validated following questionnaire :The European Organization for Research and Treatment of Cancer Breast-Cancer-Specific Quality of Life Questionnaire. See details at :https://www.eortc.be.
Questionnaire EORTC QLQ FA-12 Fatigue | At Baseline, every 12 weeks and 30 days after the last dose
  Patient reported outcomes and quality of life will be assessed using the validated following questionnaire : EORTC QLQ FA-12 Fatigue.
  The European Organisation for Research and Treatment of Cancer (EORTC) Group has developed a multidimensional instrument measuring cancer-related fatigue to be used in conjunction with the quality of life core questionnaire (EORTC QLQ-C30). The module EORTC QLQ-FA12 assesses physical, cognitive, and emotional aspects of cancer-related fatigue. See details at :https://www.eortc.be.
Questionnaire patient self-rating mood scale. | At Baseline, every 12 weeks and 30 days after the last dose
  Patient reported outcomes and quality of life will be assessed using the following questionnaire : patient self-rating mood scale.
Mutational profiles | At Baseline and in case of disease relapse up to 2 years
  To define the molecular characteristics of the tumor' patients: Mutational profiles of tumors (Whole Exome seq,)
Copy Number alterations. | At Baseline and in case of disease relapse up to 2 years
  To define the molecular characteristics of the tumor' patients: Copy Number alterations.
Loss of heterozygosity. | At Baseline and in case of disease relapse up to 2 years
  To define the molecular characteristics of the tumor' patients: loss of heterozygosity.
Circulating tumor DNA | At Baseline and in case of disease relapse up to 2 years
  Circulating tumor DNA detection and analysis will be performed on tumor' patients.
Molecular Subtyping | At Baseline and in case of disease relapse up to 2 years
  To define Molecular Subtyping of TNBC (RNAseq) on tumor' patients.
Immune monitoring | At cycle1 (each cycle is 21 days), cycle 2, cycle 5 and 24 months after randomisation or in case of relapse
  To perform Immune monitoring of circulating immune cells and circulating tumor cells on blood sample.
Circulating growth factors | At cycle1 (each cycle is 21 days), cycle 2, cycle 5 and 24 months after randomisation or in case of relapse
  To assess levels of circulating growth factors and cytokines on blood sample.
Cytokines | At cycle1 (each cycle is 21 days), cycle 2, cycle 5 and 24 months after randomisation or in case of relapse
  To assess levels of cytokines on blood sample.
PDL1 | At cycle1 (each cycle is 21 days), cycle 2, cycle 5 and 24 months after randomisation or in case of relapse
  To assess the presence in plasma of soluble PDL1.
PDL2 | At cycle1 (each cycle is 21 days), cycle 2, cycle 5 and 24 months after randomisation or in case of relapse
  To assess the presence in plasma of soluble PDL2.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Tredan, MD, Principal Investigator — Centre Leon Berard
Locations (17):
- France (17):
  - Institut de Cancérologie de l'Ouest, Angers
  - Institut Sainte Catherine, Avignon
  - CHRU Besançon, Besançon
  - Centre Francois Baclesse, Caen
  - Centre d'Oncologie Radiothérapie 37, Chambray-lès-Tours
  - Hopital Prive Jean Mermoz, Lyon
  - Centre Léon Bérard, Lyon
  - Clinique de la Sauvegarde, Lyon
  - Institut Paoli Calmettes, Marseille
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - GH Pitié-Salpêtrière-Charles Foix, Paris
  - Institut Jean Godinot, Reims
  - Institut Curie, Saint-Cloud
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Centre Paul Strauss, Strasbourg
  - Hôpital Drôme Ardèche, Valence

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tredan O, Loirat D, Chabaud S, Toussaint P, Petit T, Viret F, Levy C, Robert A, Grenier J, Mansi L, Spano JP, Patsouris A, Derbel O, Jouannaud C, Ferrero JM, Frenel JS, Molin Y, Doublet L, Heudel PE, Pierga JY, Garin G, Perol D, Bachelot T. Nivolumab in combination with ipilimumab versus capecitabine as post-operative treatment for triple negative breast cancer patients with residual disease after neoadjuvant chemotherapy: a multicentre, randomized, open-label phase II trial - BREASTIMMUNE-03. Breast. 2025 Nov 21;85:104648. doi: 10.1016/j.breast.2025.104648. Online ahead of print. PMID 41314029